CLINICAL TRIAL: NCT02835326
Title: The Collaborative Lifestyle Intervention Program in Knee Osteoarthritis Patients: CLIP-OA
Brief Title: Collaborative Lifestyle Intervention Program in Knee Osteoarthritis Patients
Acronym: CLIP-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Brian Focht, Associate Chair, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015H0394; R01AG050725 (NIH)
Record Dates: First submitted 2016-07-13; First posted 2016-07-18 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis
Keywords: Older Adults; Weight Loss; Exercise; Knee pain
MeSH Terms: conditions — Osteoarthritis; Weight Loss; Motor Activity | interventions — Exercise; Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and Dietary Weight Loss (Experimental): For the first 6 months, participants will meet at a community center for 3 group-based sessions and 1 individual session each month. Sessions include a 45 minute exercise component and a 45 minute dietary weight loss component. Exercise will consist of progressive aerobic and strength training. The dietary component will focus on decreasing caloric intake, while being nutritionally safe. All diets will be monitored by a Registered Dietitian. During months 7-12, participants will meet for 1 group session and 1 individual session per month. The final 12-24 months, bimonthly phone calls are provided to the participants to aid in retention efforts.
  Interventions: Behavioral: Exercise and Dietary Weight Loss
- Walk with Ease (Active Comparator): The Arthritis Foundation's (AF) WWE is a self-management program for symptoms of arthritis (pain, fatigue, stiffness,etc.) through exercise. It is a 6 week program involving 3 sessions per week each lasting about 60 minutes. The WWE sessions are comprised of walking, stretching and strengthening exercises, and health education lectures. These group classes will be lead by an AF instructor. Each participant will complete 2 consecutive WWE classes for a total of 12 weeks in the program. During the final week of the program, participants will be trained and transitioin to the self-directed version of WWE for maintenance of exercise. To aid in retention efforts, phone contacts are provided to participants on a monthly basis from 4-12 months and bi-monthly from 12 to 24 months
  Interventions: Behavioral: Walk with Ease

INTERVENTIONS:
Behavioral: Exercise and Dietary Weight Loss — The EX+DWL intervention consists of group and individual exercise sessions, as well as, nutritional and dietary counseling. Bimonthly phone calls are made in the final year of the study to aid in maintenance of the program.
  Arms: Exercise and Dietary Weight Loss
Behavioral: Walk with Ease — The WWE 6 week program consists of health education lectures on arthritis self-management, a walking exercise portion, and at- home strength exercises. Participants will complete two consecutive WWE programs. Monthly and bimonthly phone calls are made to participants in months 4-12 and 12-24, respectively, to aid in maintenance of the program.
  Arms: Walk with Ease

SUMMARY:
The Collaborative Lifestyle Intervention Program in Knee OsteoArthritis Patients (CLIP-OA) compares a novel community-based exercise and dietary weight loss program to the Arthritis Foundation's Walk with Ease intervention on improved mobility in knee osteoarthritis (OA) patients.

DETAILED DESCRIPTION:
Knee OA is a chronic, progressive, degenerative disease that affects over 20 million Americans, and is cited as the primary cause for activity restriction and physical disability in older adults. The joint damage and symptoms (i.e., pain, stiffness, and fatigue) accompanying symptomatic knee OA result in activity restriction, muscle atrophy, reduced quality of life and difficulty in performance of functional tasks.

Despite the well-established benefits of the Arthritis Foundation's (AF) exercise programs, recent evidence suggests that lifestyle interventions combining Exercise and Dietary Weight Loss (EX+DWL) results in superior improvements in key clinical outcomes in older, overweight or obese knee OA patients.

Primary Aim: To compare the effects of a novel community-based EX+DWL program to AF's Walk with Ease (WWE) EX intervention on improved mobility in knee osteoarthritis (OA) patients.

Secondary Aim: To compare the cost effectiveness and effects of the EX+DWL and WWE interventions on weight loss, pain, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee OA: physician documented radiographic tibiofemoral OA of one or both knees
* Overweight or Obese: BMI >25 and <40
* Knee Pain and Risk for Mobility Disability: self-reported difficulty walking ¼ mile, climbing stairs, lifting or carrying groceries, or performing other household activities due to knee pain
* Sedentary: sedentary lifestyle defined as currently participating < 20 minutes of weekly structured moderate intensity exercise occurring in bouts >10 min
* Health Status: all participants must be free of severe heart or systemic disease that would make moderate intensity exercise participation unsafe
* Age: > 50 years of age
* Stability of Residence: does not plan to move out of the Columbus metropolitan area for the duration of the study
* Consents: willing to give an informed consent and sign a HIPPA authorization form; (9) Physician Consent: treating rheumatologist and primary care physician provide medical consent for participation
* Agreeableness: willing to accept randomization and complete all assessment and intervention procedures

Exclusion Criteria:

* Health Status: any serious medical condition that precludes safe participation in an exercise program
* Study Staff Judgment: Inability to complete the study protocol, in the opinion of the study staff, due to frailty, illness, or other reasons

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-10; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Mobility Disability | baseline up to 2 years
  This will be assessed using the 400 meter walk test (400MWT), which is the time to complete 400m as quickly as possible (without running)

SECONDARY OUTCOMES:
Anthropometric Battery | baseline up to 2 years
  Body weight and height are used to calculate Body Mass Index (BMI). Body composition will be assessed using DEXA scans.
Functional Battery and Limitations | baseline up to 2 years
  Stair-climb time (SCT) is a functional performance measure that involves ascending and descending a flight of 5 stairs as quickly as possible. Limitations will be assessed using the Pepper Assessment Tool for Disability.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline up to two years
  Scale of 0 (none) to 4 (extreme) indicating the amount of difficulty they have experienced performing basic physical function tasks in the past 48 hours due to knee OA. The physical function subscale consists of 17 items that will be summed to produce a physical function score. Higher scores indicating poorer function
Rand Medical Outcomes Study 36-item Short Form Health Survey (SF-36) | baseline up to two years
  Health related quality of life survey consisting of mental and physical health with subscales of physical functioning, mental health, role-physical, role-emotional, bodily pain, general health, vitality, and social functioning
Dietary intake | baseline up to two years
  Dietary intake will be assessed by a registered dietician using the Daily food record measure. One weekend and 2 weekdays will be assessed.
Social Cognitive Process Measures | baseline up to two years
  Physical activity barriers self-efficacy scale, Satisfaction with function and appearance scale, Multiple exercise self-regulatory self-efficacy scale, the weight efficacy lifestyle questionnaire (WEL), goal commitment and goal difficulty, arthritis self-efficacy, and pain acceptance.
Change in physical activity | baseline up to two years
  Physical activity will be assessed using the Community Healthy Activities Model Program For Seniors (CHAMPS) and Lifecorder EX Accelerometer
Cost effectiveness | baseline up to two years
  The cost-effectiveness of the EX+DWL intervention compared to the WWE [program will be calculated as the ratio of additional cost per participant per increment of effectiveness. Effectiveness is based on improvement in the 400 MWT and the Quality of Well-being Scale- Self Administered (to calculate the Quality Adjusted Life Years).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Focht, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Focht BC, Rejeski WJ, Hackshaw K, Ambrosius WT, Groessl E, Chaplow ZL, DeScenza VR, Bowman J, Fairman CM, Nesbit B, Dispennette K, Zhang X, Fowler M, Haynam M, Hohn S. The Collaborative Lifestyle Intervention Program in Knee Osteoarthritis Patients (CLIP-OA) trial: Design and methods. Contemp Clin Trials. 2022 Apr;115:106730. doi: 10.1016/j.cct.2022.106730. Epub 2022 Mar 11. PMID 35283261